CLINICAL TRIAL: NCT01784497
Title: Health Related Quality of Life Assessment In Egyptian Recipients After Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: PostTransplant Quality of life
Record Dates: First submitted 2013-02-02; First posted 2013-02-06 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Health Related Quality of Life
Keywords: Health Related Quality of Life (HRQL); Living Donor Liver Transplantation(LDLT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Recipients of Living Donor Liver Transplantation: Patients who will undergo Living Donor Liver Transplantation (LDLT) In Ain Shams Center For Organ Transplantation (ASCOT) .

SUMMARY:
Health Related Quality of Life Assessment In Egyptian Recipients After Living Donor Liver Transplantation

DETAILED DESCRIPTION:
This Study Aims to Evaluate:-

1. Quality of life after LDLT In Egyptian patients using short form 36 (SF - 36) score.
2. Impact of post transplant medical and psychiatric complications on quality of life

ELIGIBILITY:
Inclusion Criteria:

* Adult Egyptian patients
* 18-60 years old
* Patients transplanted for HCV related disease and /or HCC
* Informed consent

Exclusion Criteria:

* Other etiologies for end stage liver disease (such as HBV and cholestatic liver disease and autoimmune hepatitis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who will undergo LDLT In Ain Shams Center For Organ Transplantation (ASCOT) in the next 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Quality of life after LDLT In Egyptian patients using short form 36 (SF - 36) score. | 6 months

SECONDARY OUTCOMES:
Impact of post transplant medical and psychiatric complications on quality of life | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Center For Organ Transplantation (ASCOT),Ain Shams university, Cairo, Egypt